CLINICAL TRIAL: NCT07322536
Title: The Impact of Interactive Virtual Reality Training Using Haptic Gloves on Intensive Care Nurses' Aspiration Skills and Care Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ela YILMAZ COŞKUN (Other)
Responsible Party: Sponsor-Investigator, Ela YILMAZ COŞKUN, Assistant Professor, Namik Kemal University
Organization: Namik Kemal University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 168264
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Nursing Caries; Intensive Care Nursing; Aspiration; Virtual Reality
Keywords: Aspiration; Nursing; ICU; Simulation; Skills

STUDY DESIGN:
Intervention Model Description: articipants were randomly assigned to either an experimental group or a control group. Both groups were followed in parallel throughout the study period, with the experimental group receiving haptic glove-based virtual reality training and the control group receiving standard mannequin-based aspiration training.
Masking Description: This study was conducted as an open-label trial because the nature of the educational interventions (haptic glove-based virtual reality training versus standard mannequin-based training) did not allow blinding of participants or investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The nurses used haptic glove-assisted virtual reality simulation technology under the guidance of the researcher. The practice and evaluation procedures were carried out in the same manner as in the control group, including individual sessions, checklist-based assessment, a debriefing session, and the post-test administered two weeks later.
  Interventions: Behavioral: Haptic Glove-Based Virtual Reality Training
- Control Group (No Intervention): The nurses watched a demonstration video and practiced the procedure individually in the skills laboratory. Each nurse's performance was evaluated by the researcher using the Aspiration Skill Checklist. A debriefing session was then conducted, and the knowledge test was re-administered two weeks later.

INTERVENTIONS:
Behavioral: Haptic Glove-Based Virtual Reality Training — Interactive VR simulation supported by haptic gloves for aspiration training.
  Arms: Experimental Group

SUMMARY:
This randomized controlled trial examined the effect of haptic glove-based virtual reality (VR) training on the aspiration skills and caregiving behaviors of intensive care nurses. A total of 60 nurses were randomly assigned to an experimental group receiving VR simulation supported by haptic gloves or a control group receiving standard mannequin-based training. Data were collected using the Nurse Information Form, Aspiration Skill Checklist, and Caregiving Behavior Scale. While VR training was effective in supporting aspiration skill development, no statistically significant differences were found between groups in total caregiving behavior scores or its subdimensions. These findings suggest that although VR and haptic technologies are valuable for enhancing technical skills, improvements in caregiving behaviors may require longer-term or repeated educational interventions.

DETAILED DESCRIPTION:
Aspiration is a fundamental nursing intervention in intensive care units and requires advanced psychomotor skills, strict adherence to infection control principles, and consistent caregiving behaviors. Conventional training methods, such as mannequin-based demonstrations, may be limited in providing sufficient hands-on practice and realistic feedback, particularly for complex clinical procedures. Recent advances in virtual reality (VR) technology, especially systems supported by haptic gloves, offer immersive learning environments that enable repeated practice with real-time tactile feedback, potentially enhancing clinical skill acquisition.

This randomized controlled trial was conducted to determine the effect of haptic glove-based virtual reality training on the aspiration skills and caregiving behaviors of intensive care nurses. The study was carried out between November 2024 and January 2025 in the adult intensive care, coronary intensive care, and neonatal intensive care units of a foundation university hospital.

A total of 60 intensive care nurses were randomly assigned to either an experimental group or a control group. The control group received standard aspiration training using mannequin-based demonstration, while the experimental group participated in an interactive virtual reality simulation supported by haptic gloves. The VR training allowed participants to perform aspiration procedures in a simulated intensive care environment with tactile feedback, emphasizing correct procedural steps, patient safety, and evidence-based care principles.

Data were collected through face-to-face surveys using the Nurse Information Form, the Aspiration Skill Checklist, and the Caregiving Behavior Scale. Aspiration skills and caregiving behaviors were assessed before and after the training interventions. The primary outcomes of the study were aspiration skill performance and caregiving behavior scores, including the subdimensions of assurance, knowledge-skill, respectfulness, and commitment.

The findings demonstrated no statistically significant differences between the experimental and control groups in total caregiving behavior scores or in any of the caregiving behavior subdimensions. While VR-based training did not show a direct effect on caregiving behaviors, previous evidence suggests that VR and haptic technologies are particularly effective in improving technical and psychomotor skills. Behavioral and attitudinal changes may require longer-term or repeated training interventions.

The results of this study are expected to contribute to the growing body of evidence on technology-enhanced learning in nursing education and to inform the integration of haptic glove-supported virtual reality applications into intensive care nursing skills training programs.

ELIGIBILITY:
Inclusion Criteria: The inclusion criteria were as follows: being 18 years of age or older, working as an intensive care nurse and having prior experience with the aspiration procedure, being computer literate, and having no visual or hearing impairments.

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Aspiration skill performance score | Baseline (pre-test) and 2 weeks after training (post-test).
  Measured with the Aspiration Skill Checklist

SECONDARY OUTCOMES:
Caregiving behavior total and subdimension scores | Baseline and 2 weeks post-training.
  Measured with the Caregiving Behavior Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet KIZIL, PhD, Principal Investigator — Hamidiye Faculty Nursing
Locations (1):
- İstanbul Beykent University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No